CLINICAL TRIAL: NCT04386135
Title: DESVELA Cohort. Analysis of the Role of Personal Skills as Determinants of Incidence of Morbidity, Lifestyles, Quality of Life, Use of Services and Mortality.
Brief Title: DESVELA. Personal Skills as Determinants of Morbidity, Lifestyles, Quality of Life, Use of Services and Mortality.
Acronym: DESVELA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Preventive Services and Health Promotion Research Network (Other); Instituto de Salud Carlos III (Other Government); Parc Sanitari Sant Joan de Déu (Other); Servei de Salut de les Illes Balears (Unknown); Institut Català de la Salut (Other); Servicio Aragones De Salud (Other); Osakidetza (Other); Andaluz Health Service (Other Government); Castilla-La Mancha Health Service (Other); Biobizkaia Health Research Institute (Other Government); Fundació Sant Joan de Déu (Other); Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other); Universidad Loyola Andalucia (Other); University of Castilla-La Mancha (Other); Instituto de Investigación Sanitaria Aragón (Other); Fundació d'investigació Sanitària de les Illes Balears (Other Government); Fundacin Biomedica Galicia Sur (Other); Public Health Service of Galicia (Other)
Responsible Party: Sponsor
Other Study IDs: 4R19/112; PI19/01285 (Other Grant/Funding Number: Instituto de Salud Carlos III.); PI19/00147 (Other Grant/Funding Number: Instituto de Salud Carlos III.); PI19/01459 (Other Grant/Funding Number: Instituto de Salud Carlos III.); PI19/00997 (Other Grant/Funding Number: Instituto de Salud Carlos III.); PI19/00115 (Other Grant/Funding Number: Instituto de Salud Carlos III.); PI19/01140 (Other Grant/Funding Number: Instituto de Salud Carlos III.); PI19/01264 (Other Grant/Funding Number: Instituto de Salud Carlos III.); PI19/00434 (Other Grant/Funding Number: Instituto de Salud Carlos III.); PI19/01314 (Other Grant/Funding Number: Instituto de Salud Carlos III.); PI19/01076 (Other Grant/Funding Number: Instituto de Salud Carlos III.)
Record Dates: First submitted 2020-04-30; First posted 2020-05-13 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: General Population; Health Knowledge, Attitudes, Practice; Empowerment; Health Care Utilization; Life Style; Self Efficacy; Activation, Patient; Locus of Control; Quality of Life
Keywords: Primary Health Care; Health Promotion; Quality of Life; Life Style; Health Literacy; Empowerment; Locus of Control; Personality; Self Efficacy
MeSH Terms: conditions — Behavior; Empowerment; Patient Acceptance of Health Care; Patient Participation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Quantitative study: The main objective is to analyze whether personal skills related to behaviours are independently associated with the incidence of morbidity. Study with quantitative and qualitative methodology. Multicenter project (10 teams) for the creation of a cohort of 3083 people aged 35 to 74 years of 9 Autonomous Communities (AACC). The personal variables that will be evaluated are: self-efficacy, activation, health literacy, resilience, locus of control and personality traits. Socio-demographic covariates, social capital and community health assets will be recorded. As a secondary objective, it will be analyzed whether personal skills are independently associated with lower all cause mortality, better adoption of healthy lifestyles, higher quality of life and less utilization of health services in follow-up. A physical examination, a blood analytical and a cognitive evaluation will be carried out. The incidence of morbidity will be analyzed with a Cox model for each of the six independent variables (objective 1); and mortality from all causes and from the other dependent variables (objective 2). The models will be adjusted by the indicated covariables. The possible heterogeneity between (AACC) will be estimated by introducing random effects into the model.

Qualitative study: To deepen in the opinions and experiences of the population on the relationship between personal skills with their perception of health, their lifestyles and their quality of life. The research will be carried out from a phenomenological perspective. The number of discussion groups needed to reach the saturation of speeches will be made. There will be an analysis of thematic content that will be triangulated between members of the research team. The meanings will be interpreted and an explanatory framework will be created with the contributions of each type of informant.

ELIGIBILITY:
Inclusion Criteria:

- Population ascribed to Primary Health Centres in Spain.

Exclusion Criteria:

* Illness at terminal phase.
* Institutionalization.
* Intellectual disability.
* Dementia.
* Idiomatic difficulties

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population adscrited to Primary Health Centres in Spain
Sampling Method: Probability Sample
Enrollment: 3260 (Actual)
Dates: Start 2021-06-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of morbidity. | Five years
  The following pathologies will be considered in the evaluation of morbidity. 1) hypertension (HTA) 2) ischemic heart disease 3) heart failure 4) cardiac arrhythmias 5) diabetes mellitus (DM) 6) ischemic stroke 7) peripheral artery disease (PAD) 8) chronic obstructive pulmonary disease 9) asthma 10) any type of arthritis 11) osteoporosis 12) any type of cancer 13) Parkinson's disease 14) affective disorders 15) psychotic disorders 16) dementia 17) obesity. The appearance of a new condition in the clinical health history (CHI) in the follow-up, in relation to the ones it had in the baseline, will be considered. But in 4 cases, information of the physical exploration will be also considered. - HTA: in CHI or treatment for hypertension or systolic blood pressure ≥140 mmHg or Diastolic BP ≥90 mmHg. - DM: in CHI or treatment for diabetes or fasting glucose ≥ 126 mg/dL. - PAD: in CHI or ankle-brachial index <0.9.- Obesity: in CHI or body mass index: weight/ height2 is ≥30 kg/m2.
Incidence of morbidity. | Ten years
  The following pathologies will be considered in the evaluation of morbidity. 1) hypertension (HTA) 2) ischemic heart disease 3) heart failure 4) cardiac arrhythmias 5) diabetes mellitus (DM) 6) ischemic stroke 7) peripheral artery disease (PAD) 8) chronic obstructive pulmonary disease 9) asthma 10) any type of arthritis 11) osteoporosis 12) any type of cancer 13) Parkinson's disease 14) affective disorders 15) psychotic disorders 16) dementia 17) obesity. The appearance of a new condition in the clinical health history (CHI) in the follow-up, in relation to the ones it had in the baseline, will be considered. But in 4 cases, information of the physical exploration will be also considered. - HTA: in CHI or treatment for hypertension or systolic blood pressure ≥140 mmHg or Diastolic BP ≥90 mmHg. - DM: in CHI or treatment for diabetes or fasting glucose ≥ 126 mg/dL. - PAD: in CHI or ankle-brachial index <0.9.- Obesity: in CHI or body mass index: weight/ height2 is ≥30 kg/m2.
Mortality from all causes | Five years
  Mortality and its causes will be known by checking health care records.
Mortality from all causes | Ten years
  Mortality and its causes will be known by checking health care records.
Self-reported adherence to Mediterranean diet (PREDIMED scale) | Five years
  The questionnaire is validated in Spain in Spanish. Adherence to Mediterranean diet (PREDIMED; 0-14, higher values = higher adherence; ref: Martínez-González MA et al. (2012). PLoS One 7:e43134)
Self-reported adherence to Mediterranean diet (PREDIMED scale) | Ten years
  The questionnaire is validated in Spain in Spanish. Adherence to Mediterranean diet (PREDIMED; 0-14, higher values = higher adherence; ref: Martínez-González MA et al. (2012). PLoS One 7:e43134)
Self-reported physical activity (Validated questionnaire) | Five years
  Level of physical activity (higher score = higher level of PA, Physical activity expenditure is estimated in metabolic equivalent of task (MET) METs-hour-week; ref: Puig-Ribera A, et al. (2015). PLoS One 10:e0136870);
Self-reported physical activity (Validated questionnaire) | Ten years
  Level of physical activity (higher score = higher level of PA, Physical activity expenditure is estimated in METs-hour-week; ref: Puig-Ribera A, et al. (2015). PLoS One 10:e0136870);
Tobacco Consumption | Five years
  Tobacco consumption, 4-question scale adapted from the World Health Organization (WHO) MONICA Study
Tobacco Consumption | Ten years
  Tobacco consumption, 4-question scale adapted from the WHO MONICA Study
Alcohol consumption | Five years
  Alcohol consumption, will be assessed by self-reported units during the last week, and a question regarding the monthly frequency during the last year of excessive alcohol consumption (alcohol binge drinking)
Alcohol consumption | Ten years
  Alcohol consumption, will be assessed by self-reported units during the last week, and a question regarding the monthly frequency during the last year of excessive alcohol consumption (alcohol binge drinking)
Insomnia assessment | Five years
  Insomnia will be measured with the Pittsburgh Sleep Quality Index (PSQI); 0-21, Higher scores represent poorer subjective sleep quality; ref: Hita-Contreras, F. et al. (2014). Rheumatology International, 34(7), 929-936).
Insomnia assessment | Ten years
  Insomnia will be measured with the Pittsburgh Sleep Quality Index-PSQI; 0-21, Higher scores represent poorer subjective sleep quality; ref: Hita-Contreras, F. et al. (2014). Rheumatology International, 34(7), 929-936).
Self-reported quality of of life | Five years
  Quality of life will be measured with EuroQol5D (number of dimensions with problems) + EVA (0-100, higher value higher perception of quality of life); ref: Herdman M, et al. (2015). Aten Primaria 28(6): 425-9).
Self-reported quality of of life | Ten years
  Quality of life will be measured with EuroQol 5D (number of dimensions with problems) + visual analogue scale (VAS) (0-100, higher value higher perception of quality of life); ref: Herdman M, et al. (2015). Aten Primaria 28(6): 425-9).
Health service use | Five years
  Use of health services will be recorded from the health electronic records of each participant.
Health service use | Ten years
  Use of health services will be recorded from the health electronic records of each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventura Bolíbar, Study Chair — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina; Rafel Ramos, PhD, Study Director — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina; Ruth Martí-Lluch, PhD, Principal Investigator — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Locations (20):
- Spain (20):
  - Centro de Salud Olivar de Quintos., Dos Hermanas, Andalusia
  - Centro de Salud de Ferreries, Bisbe Severo, 3., Ferreries, Balearic Islands
  - Centro de Salud de Manacor, C/d'En Simó Tort, 19., Manacor, Balearic Islands
  - CAP Cornellà SDPI, La Gavarra. Carrer de Bellaterra, 41., Cornellà de Llobregat, Barcelona
  - CAP Sant Ildefons. Avinguda de la República Argentina, S/N., Cornellà de Llobregat, Barcelona
  - CAP Dr. Bartomeu Fabrés Anglada Gava 2. Carrer de la Riera de les Parets, 7., Gavà, Barcelona
  - CAP Alhambra. Carrer de l'Alhambra, 20., L'Hospitalet de Llobregat, Barcelona
  - Centro de Salud de Deusto, Luis Power, 18., Bilbao, Bizkaia
  - Centro de Salud de Leiro, C/Gabino Bugallal S/N., Leiro, Orense
  - Centro de Salud Beiramar, AV. da Beiramar, 51., Vigo, Pontevedra
  - Centro de Salud Guijuelo. C/ Teso de La Feria, S/N., Guijuelo, Salamanca
  - Centro de Salud Linares de Riofrío. Ctra. de Guijuelo, S/N., Linares de Riofrío, Salamanca
  - Centro de Salud Peñafiel. Carrer Cruz Roja, S/N., Peñafiel, Valladolid
  - Centro de Salud Tudela de Duero. C/ María Zambrano, S/N., Tudela de Duero, Valladolid
  - Centro de Salud San Pablo. C/ Cardenal Torquemada, S/N., Valladolid, Valladolid
  - CS Daroca. C/Luchente S/N, Daroca, Zaragoza
  - Centro de Salud Cuenca 1, Calle Colón 2., Cuenca
  - Unidad de Investigación en Atención Primaria de Girona, IDIAP Jordi Gol, Institut Català de la Salut, Girona
  - Centro de Salud San Juan. Avda. de Portugal, 83-89., Salamanca
  - CS Arrabal, C/Andador Aragüés del Puerto, 3., Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mounce LTA, Campbell JL, Henley WE, Tejerina Arreal MC, Porter I, Valderas JM. Predicting Incident Multimorbidity. Ann Fam Med. 2018 Jul;16(4):322-329. doi: 10.1370/afm.2271. PMID 29987080
- [Background] Noncommunicable diseases country profiles 2018. Geneva: World Health Organization; 2018. Licence CC BY-NC-SA 3.0 IGO.
- [Background] World Health Organization (WHO). Global status report on noncommunicable diseases 2014. Ginebra; 2014. ISBN 978 92 4 156422 8. [Internet]. Disponible en: http://www.who.int/nmh/publications/ncd_report_full_en.pdf.
- [Background] Kessler RC, Aguilar-Gaxiola S, Alonso J, Chatterji S, Lee S, Ormel J, Ustun TB, Wang PS. The global burden of mental disorders: an update from the WHO World Mental Health (WMH) surveys. Epidemiol Psichiatr Soc. 2009 Jan-Mar;18(1):23-33. doi: 10.1017/s1121189x00001421. PMID 19378696
- [Background] O'Neil A, Jacka FN, Quirk SE, Cocker F, Taylor CB, Oldenburg B, Berk M. A shared framework for the common mental disorders and Non-Communicable Disease: key considerations for disease prevention and control. BMC Psychiatry. 2015 Feb 5;15:15. doi: 10.1186/s12888-015-0394-0. PMID 25652365
- [Background] Carta de Ottawa para la Promoción de la Salud, OMS, Ginebra, 1986. Who.int. (2015). WHO. [internet] Disponible en: http://www.who.int/healthpromotion/conferences/previous/ottawa/en/index1.html.
- [Background] Gol i Gurina J. Els Grans Temes D'un Pensament I D'una Vida. Barcelona: La llar del llibre; 1986
- [Background] Rosenzveig A, Kuspinar A, Daskalopoulou SS, Mayo NE. Toward patient-centered care: a systematic review of how to ask questions that matter to patients. Medicine (Baltimore). 2014 Nov;93(22):e120. doi: 10.1097/MD.0000000000000120. PMID 25396331
- [Background] Declaración de Yakarta, YAkarta, 1997. WHO. [internet] Disponible en: http://www.who.int/healthpromotion/conferences/previous/jakarta/en/hpr_jakarta_declaration_sp.pdf
- [Background] Estrategia de promoción de la salud y prevención en el SNS. Madrid, 2013. MSSSI. Disponible en: https://www.msssi.gob.es/profesionales/saludPublica/prevPromocion/Estrategia/estrategiaPromocionyPrevencion.htm
- [Background] Dahlgren G, Whitehead M. Policies and strategies to promote social equity in health. Stockholm: Institute for future studies; 1991. [internet]. Disponible en: https://core.ac.uk/download/pdf/6472456.pdf.
- [Background] Antonovsky A. The salutogenic model as a theory to guide health promotion. Health Promotion International. 1996;11:11-18.
- [Background] Marmot M. 2004. The Status Syndrome: How Social Standing Affects Our Health and Longevity. New York: Henry Holt.
- [Background] Atkins L, Francis J, Islam R, O'Connor D, Patey A, Ivers N, Foy R, Duncan EM, Colquhoun H, Grimshaw JM, Lawton R, Michie S. A guide to using the Theoretical Domains Framework of behaviour change to investigate implementation problems. Implement Sci. 2017 Jun 21;12(1):77. doi: 10.1186/s13012-017-0605-9. PMID 28637486
- [Background] Rammstedt B, John OP. Measuring personality in one minute or less: A 10-item short version of the Big Five Inventory in English and German. J Res Pers. 2007; 41:203 -12.
- [Background] Goodwin RD, Friedman HS. Health status and the five-factor personality traits in a nationally representative sample. J Health Psychol. 2006 Sep;11(5):643-54. doi: 10.1177/1359105306066610. PMID 16908463
- [Background] Chapman BP, Fiscella K, Kawachi I, Duberstein PR. Personality, socioeconomic status, and all-cause mortality in the United States. Am J Epidemiol. 2010 Jan 1;171(1):83-92. doi: 10.1093/aje/kwp323. Epub 2009 Dec 4. PMID 19965888
- [Background] Jokela M, Pulkki-Raback L, Elovainio M, Kivimaki M. Personality traits as risk factors for stroke and coronary heart disease mortality: pooled analysis of three cohort studies. J Behav Med. 2014 Oct;37(5):881-9. doi: 10.1007/s10865-013-9548-z. Epub 2013 Nov 8. PMID 24203126
- [Background] Jokela M, Batty GD, Nyberg ST, Virtanen M, Nabi H, Singh-Manoux A, Kivimaki M. Personality and all-cause mortality: individual-participant meta-analysis of 3,947 deaths in 76,150 adults. Am J Epidemiol. 2013 Sep 1;178(5):667-75. doi: 10.1093/aje/kwt170. Epub 2013 Aug 1. PMID 23911610
- [Background] Hengartner MP, Kawohl W, Haker H, Rossler W, Ajdacic-Gross V. Big Five personality traits may inform public health policy and preventive medicine: Evidence from a cross-sectional and a prospective longitudinal epidemiologic study in a Swiss community. J Psychosom Res. 2016 May;84:44-51. doi: 10.1016/j.jpsychores.2016.03.012. Epub 2016 Mar 24. PMID 27095158
- [Background] Rotter JB. Generalized expectancies for internal versus external control of reinforcement. Psychol Monogr. 1966;80(1):1-28. No abstract available. PMID 5340840
- [Background] Berglund E, Lytsy P, Westerling R. The influence of locus of control on self-rated health in context of chronic disease: a structural equation modeling approach in a cross sectional study. BMC Public Health. 2014 May 23;14:492. doi: 10.1186/1471-2458-14-492. PMID 24885619
- [Background] Sturmer T, Hasselbach P, Amelang M. Personality, lifestyle, and risk of cardiovascular disease and cancer: follow-up of population based cohort. BMJ. 2006 Jun 10;332(7554):1359. doi: 10.1136/bmj.38833.479560.80. Epub 2006 May 10. PMID 16687457
- [Background] Moreno-Peral P, Conejo-Ceron S, Fernandez A, Berenguera A, Martinez-Andres M, Pons-Vigues M, Motrico E, Rodriguez-Martin B, Bellon JA, Rubio-Valera M. Primary care patients' perspectives of barriers and enablers of primary prevention and health promotion-a meta-ethnographic synthesis. PLoS One. 2015 May 4;10(5):e0125004. doi: 10.1371/journal.pone.0125004. eCollection 2015. PMID 25938509
- [Background] Wilski M, Chmielewski B, Tomczak M. Work locus of control and burnout in Polish physiotherapists: The mediating effect of coping styles. Int J Occup Med Environ Health. 2015;28(5):875-89. doi: 10.13075/ijomeh.1896.00287. PMID 26224499
- [Background] Poortinga W, Dunstan FD, Fone DL. Health locus of control beliefs and socio-economic differences in self-rated health. Prev Med. 2008 Apr;46(4):374-80. doi: 10.1016/j.ypmed.2007.11.015. Epub 2007 Dec 4. PMID 18177930
- [Background] Mautner D, Peterson B, Cunningham A, Ku B, Scott K, LaNoue M. How Multidimensional Health Locus of Control predicts utilization of emergency and inpatient hospital services. J Health Psychol. 2017 Mar;22(3):314-323. doi: 10.1177/1359105315603468. Epub 2016 Jul 10. PMID 26430065
- [Background] Henninger DE, Whitson HE, Cohen HJ, Ariely D. Higher medical morbidity burden is associated with external locus of control. J Am Geriatr Soc. 2012 Apr;60(4):751-5. doi: 10.1111/j.1532-5415.2012.03904.x. Epub 2012 Mar 28. PMID 22458257
- [Background] Keedy NH, Keffala VJ, Altmaier EM, Chen JJ. Health locus of control and self-efficacy predict back pain rehabilitation outcomes. Iowa Orthop J. 2014;34:158-65. PMID 25328476
- [Background] Sherer M, Maddux JE, Mercandante B, Prentice-Dunn S, Jacobs B, Rogers RW. The Self-Efficacy Scale: Construction and Validation. Psychol Rep. 1982;51:663 -71.
- [Background] Groffen DA, Bosma H, Tan FE, van den Akker M, Kempen GI, van Eijk JT. Material vs. psychosocial explanations of old-age educational differences in physical and mental functioning. Eur J Public Health. 2012 Aug;22(4):587-92. doi: 10.1093/eurpub/ckr063. Epub 2011 Jun 6. PMID 21646362
- [Background] Windsor TD, Anstey KJ. A longitudinal investigation of perceived control and cognitive performance in young, midlife and older adults. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2008 Nov;15(6):744-63. doi: 10.1080/13825580802348570. Epub 2008 Sep 11. PMID 18787982
- [Background] Zahodne LB, Nowinski CJ, Gershon RC, Manly JJ. Which psychosocial factors best predict cognitive performance in older adults? J Int Neuropsychol Soc. 2014 May;20(5):487-95. doi: 10.1017/S1355617714000186. Epub 2014 Mar 31. PMID 24685143
- [Background] Bardach SH, Schoenberg NE, Howell BM. What Motivates Older Adults to Improve Diet and Exercise Patterns? J Community Health. 2016 Feb;41(1):22-9. doi: 10.1007/s10900-015-0058-5. PMID 26159781
- [Background] Olsson I, Dahl AA. Avoidant personality problems--their association with somatic and mental health, lifestyle, and social network. A community-based study. Compr Psychiatry. 2012 Aug;53(6):813-21. doi: 10.1016/j.comppsych.2011.10.007. Epub 2011 Dec 5. PMID 22146705
- [Background] Dolores Serrano-Parra M, Garrido-Abejar M, Notario-Pacheco B, Bartolome-Gutierrez R, Solera-Martinez M, Martinez-Vizcaino V. [Validity of the Connor-Davidson resilience scale (10 items) in a population of elderly]. Enferm Clin. 2013 Jan-Feb;23(1):14-21. doi: 10.1016/j.enfcli.2012.11.006. Epub 2013 Jan 23. Spanish. PMID 23352433
- [Background] Notario-Pacheco B, Solera-Martinez M, Serrano-Parra MD, Bartolome-Gutierrez R, Garcia-Campayo J, Martinez-Vizcaino V. Reliability and validity of the Spanish version of the 10-item Connor-Davidson Resilience Scale (10-item CD-RISC) in young adults. Health Qual Life Outcomes. 2011 Aug 5;9:63. doi: 10.1186/1477-7525-9-63. PMID 21819555
- [Background] Norris FH, Stevens SP, Pfefferbaum B, Wyche KF, Pfefferbaum RL. Community resilience as a metaphor, theory, set of capacities, and strategy for disaster readiness. Am J Community Psychol. 2008 Mar;41(1-2):127-50. doi: 10.1007/s10464-007-9156-6. PMID 18157631
- [Background] Davydov DM, Stewart R, Ritchie K, Chaudieu I. Resilience and mental health. Clin Psychol Rev. 2010 Jul;30(5):479-95. doi: 10.1016/j.cpr.2010.03.003. Epub 2010 Mar 25. PMID 20395025
- [Background] Lang FR, Heckhausen J. Perceived control over development and subjective well-being: differential benefits across adulthood. J Pers Soc Psychol. 2001 Sep;81(3):509-23. doi: 10.1037//0022-3514.81.3.509. PMID 11554650
- [Background] Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the Patient Activation Measure (PAM): conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004 Aug;39(4 Pt 1):1005-26. doi: 10.1111/j.1475-6773.2004.00269.x. PMID 15230939
- [Background] Vernooij RW, Willson M, Gagliardi AR; members of the Guidelines International Network Implementation Working Group. Characterizing patient-oriented tools that could be packaged with guidelines to promote self-management and guideline adoption: a meta-review. Implement Sci. 2016 Apr 14;11:52. doi: 10.1186/s13012-016-0419-1. PMID 27079375
- [Background] Blakemore A, Hann M, Howells K, Panagioti M, Sidaway M, Reeves D, Bower P. Patient activation in older people with long-term conditions and multimorbidity: correlates and change in a cohort study in the United Kingdom. BMC Health Serv Res. 2016 Oct 18;16(1):582. doi: 10.1186/s12913-016-1843-2. PMID 27756341
- [Background] Moreno-Chico C, Gonzalez-de Paz L, Monforte-Royo C, Arrighi E, Navarro-Rubio MD, Gallart Fernandez-Puebla A. Adaptation to European Spanish and psychometric properties of the Patient Activation Measure 13 in patients with chronic diseases. Fam Pract. 2017 Sep 1;34(5):627-634. doi: 10.1093/fampra/cmx022. PMID 28379415
- [Background] Sorensen K, Pelikan JM, Rothlin F, Ganahl K, Slonska Z, Doyle G, Fullam J, Kondilis B, Agrafiotis D, Uiters E, Falcon M, Mensing M, Tchamov K, van den Broucke S, Brand H; HLS-EU Consortium. Health literacy in Europe: comparative results of the European health literacy survey (HLS-EU). Eur J Public Health. 2015 Dec;25(6):1053-8. doi: 10.1093/eurpub/ckv043. Epub 2015 Apr 5. PMID 25843827
- [Background] Dewalt DA, Berkman ND, Sheridan S, Lohr KN, Pignone MP. Literacy and health outcomes: a systematic review of the literature. J Gen Intern Med. 2004 Dec;19(12):1228-39. doi: 10.1111/j.1525-1497.2004.40153.x. PMID 15610334
- [Background] Dennis S, Williams A, Taggart J, Newall A, Denney-Wilson E, Zwar N, Shortus T, Harris MF. Which providers can bridge the health literacy gap in lifestyle risk factor modification education: a systematic review and narrative synthesis. BMC Fam Pract. 2012 May 28;13:44. doi: 10.1186/1471-2296-13-44. PMID 22639799
- [Background] Stringhini S, Carmeli C, Jokela M, Avendano M, Muennig P, Guida F, Ricceri F, d'Errico A, Barros H, Bochud M, Chadeau-Hyam M, Clavel-Chapelon F, Costa G, Delpierre C, Fraga S, Goldberg M, Giles GG, Krogh V, Kelly-Irving M, Layte R, Lasserre AM, Marmot MG, Preisig M, Shipley MJ, Vollenweider P, Zins M, Kawachi I, Steptoe A, Mackenbach JP, Vineis P, Kivimaki M; LIFEPATH consortium. Socioeconomic status and the 25 x 25 risk factors as determinants of premature mortality: a multicohort study and meta-analysis of 1.7 million men and women. Lancet. 2017 Mar 25;389(10075):1229-1237. doi: 10.1016/S0140-6736(16)32380-7. Epub 2017 Feb 1. PMID 28159391
- [Background] Marmot M, Allen J, Bell R, Bloomer E, Goldblatt P; Consortium for the European Review of Social Determinants of Health and the Health Divide. WHO European review of social determinants of health and the health divide. Lancet. 2012 Sep 15;380(9846):1011-29. doi: 10.1016/S0140-6736(12)61228-8. Epub 2012 Sep 8. PMID 22964159
- [Background] Reblin M, Uchino BN. Social and emotional support and its implication for health. Curr Opin Psychiatry. 2008 Mar;21(2):201-5. doi: 10.1097/YCO.0b013e3282f3ad89. PMID 18332671
- [Background] Moore S, Kawachi I. Twenty years of social capital and health research: a glossary. J Epidemiol Community Health. 2017 May;71(5):513-517. doi: 10.1136/jech-2016-208313. Epub 2017 Jan 13. PMID 28087811
- [Background] Villalonga-Olives E, Kawachi I. The dark side of social capital: A systematic review of the negative health effects of social capital. Soc Sci Med. 2017 Dec;194:105-127. doi: 10.1016/j.socscimed.2017.10.020. Epub 2017 Oct 21. PMID 29100136
- [Background] Poortinga W. Social relations or social capital? Individual and community health effects of bonding social capital. Soc Sci Med. 2006 Jul;63(1):255-70. doi: 10.1016/j.socscimed.2005.11.039. Epub 2006 Jan 19. PMID 16427171
- [Background] Kim D, Subramanian SV, Kawachi I. Bonding versus bridging social capital and their associations with self rated health: a multilevel analysis of 40 US communities. J Epidemiol Community Health. 2006 Feb;60(2):116-22. doi: 10.1136/jech.2005.038281. PMID 16415259
- [Background] House JS, Landis KR, Umberson D. Social relationships and health. Science. 1988 Jul 29;241(4865):540-5. doi: 10.1126/science.3399889.
- [Background] Holt-Lunstad J, Smith TB, Layton JB. Social relationships and mortality risk: a meta-analytic review. PLoS Med. 2010 Jul 27;7(7):e1000316. doi: 10.1371/journal.pmed.1000316. PMID 20668659
- [Background] Ehsan AM, De Silva MJ. Social capital and common mental disorder: a systematic review. J Epidemiol Community Health. 2015 Oct;69(10):1021-8. doi: 10.1136/jech-2015-205868. Epub 2015 Jul 15. PMID 26179447
- [Background] Siegrist J, Starke D, Chandola T, Godin I, Marmot M, Niedhammer I, Peter R. The measurement of effort-reward imbalance at work: European comparisons. Soc Sci Med. 2004 Apr;58(8):1483-99. doi: 10.1016/S0277-9536(03)00351-4. PMID 14759692
- [Background] Rugulies R, Aust B, Madsen IE, Burr H, Siegrist J, Bultmann U. Adverse psychosocial working conditions and risk of severe depressive symptoms. Do effects differ by occupational grade? Eur J Public Health. 2013 Jun;23(3):415-20. doi: 10.1093/eurpub/cks071. Epub 2012 Jun 8. PMID 22683769
- [Background] Rugulies R, Aust B, Madsen IE. Effort-reward imbalance at work and risk of depressive disorders. A systematic review and meta-analysis of prospective cohort studies. Scand J Work Environ Health. 2017 Jul 1;43(4):294-306. doi: 10.5271/sjweh.3632. Epub 2017 Mar 17. PMID 28306759
- [Background] Fahlen G, Knutsson A, Peter R, Akerstedt T, Nordin M, Alfredsson L, Westerholm P. Effort-reward imbalance, sleep disturbances and fatigue. Int Arch Occup Environ Health. 2006 May;79(5):371-8. doi: 10.1007/s00420-005-0063-6. Epub 2005 Dec 13. PMID 16362323
- [Background] Dragano N, Siegrist J, Nyberg ST, Lunau T, Fransson EI, Alfredsson L, Bjorner JB, Borritz M, Burr H, Erbel R, Fahlen G, Goldberg M, Hamer M, Heikkila K, Jockel KH, Knutsson A, Madsen IEH, Nielsen ML, Nordin M, Oksanen T, Pejtersen JH, Pentti J, Rugulies R, Salo P, Schupp J, Singh-Manoux A, Steptoe A, Theorell T, Vahtera J, Westerholm PJM, Westerlund H, Virtanen M, Zins M, Batty GD, Kivimaki M; IPD-Work consortium. Effort-Reward Imbalance at Work and Incident Coronary Heart Disease: A Multicohort Study of 90,164 Individuals. Epidemiology. 2017 Jul;28(4):619-626. doi: 10.1097/EDE.0000000000000666. PMID 28570388
- [Background] Burgel BJ, White MC, Gillen M, Krause N. Psychosocial work factors and shoulder pain in hotel room cleaners. Am J Ind Med. 2010 Jul;53(7):743-56. doi: 10.1002/ajim.20832. PMID 20340100
- [Background] Siegrist J, Li J. Work Stress and Altered Biomarkers: A Synthesis of Findings Based on the Effort-Reward Imbalance Model. Int J Environ Res Public Health. 2017 Nov 10;14(11):1373. doi: 10.3390/ijerph14111373. PMID 29125555
- [Background] Van Bortel T, Wickramasinghe ND, Morgan A, Martin S. Health assets in a global context: a systematic review of the literature. BMJ Open. 2019 Feb 3;9(2):e023810. doi: 10.1136/bmjopen-2018-023810. PMID 30782888
- [Background] Violan C, Foguet-Boreu Q, Flores-Mateo G, Salisbury C, Blom J, Freitag M, Glynn L, Muth C, Valderas JM. Prevalence, determinants and patterns of multimorbidity in primary care: a systematic review of observational studies. PLoS One. 2014 Jul 21;9(7):e102149. doi: 10.1371/journal.pone.0102149. eCollection 2014. PMID 25048354
- [Background] Le Reste JY, Nabbe P, Lingner H, Kasuba Lazic D, Assenova R, Munoz M, Sowinska A, Lygidakis C, Doerr C, Czachowski S, Argyriadou S, Valderas J, Le Floch B, Deriennic J, Jan T, Melot E, Barraine P, Odorico M, Lietard C, Van Royen P, Van Marwijk H. What research agenda could be generated from the European General Practice Research Network concept of Multimorbidity in Family Practice? BMC Fam Pract. 2015 Sep 17;16:125. doi: 10.1186/s12875-015-0337-3. PMID 26381383
- [Derived] Young-Silva Y, Berenguera A, Juvinya-Canal D, Marti-Lluch R, Arroyo-Uriarte P, Tamayo-Morales O, Marcilla-Toribio I, Elizondo-Alzola U, Mendez-Lopez F, Chela-Alvarez X, Motrico E. Exploring personal aptitudes and personality traits that, together with social determinants, shape health behaviors and conduct: a thematic analysis based on the Capability, Opportunity, Motivation and Behavior (COM-B) change system. Front Public Health. 2024 Jun 5;12:1387528. doi: 10.3389/fpubh.2024.1387528. eCollection 2024. PMID 38898892
- [Derived] Marti-Lluch R, Bolibar B, Llobera J, Maderuelo-Fernandez JA, Magallon-Botaya R, Sanchez-Perez A, Fernandez-Dominguez MJ, Motrico E, Vicens-Pons E, Notario-Pacheco B, Alves-Cabratosa L, Ramos R; DESVELA Cohort Investigators. Role of personal aptitudes as determinants of incident morbidity, lifestyles, quality of life, use of health services, and mortality (DESVELA cohort): quantitative study protocol for a prospective cohort study in a hybrid analysis. Front Public Health. 2023 Jun 22;11:1067249. doi: 10.3389/fpubh.2023.1067249. eCollection 2023. PMID 37427254
- [Derived] Young-Silva Y, Berenguera A, Jacques-Avino C, Gil-Girbau M, Arroyo-Uriarte P, Chela-Alvarez X, Ripoll J, Marti-Lluch R, Ramos R, Elizondo-Alzola U, Garcia-Martinez S, Mendez-Lopez F, Tamayo-Morales O, Martinez-Andres M, Motrico E, Gomez-Gomez I, Fernandez-Alvarez R, Juvinya-Canal D; DESVELA Cohort investigators. Role of personal aptitudes as determinants of incident morbidity, lifestyles, quality of life, use of the health services and mortality (DESVELA cohort): qualitative study protocol for a prospective cohort study in a hybrid analysis. Front Public Health. 2023 Jun 9;11:1069957. doi: 10.3389/fpubh.2023.1069957. eCollection 2023. PMID 37361167